CLINICAL TRIAL: NCT03683667
Title: Efficacy of Supplemental Protein, Delivered Alone or in Combination With Treatment for Enteric Pathogens, to Prevent Growth Faltering in Bangladeshi Infants
Brief Title: Protein Plus: Improving Infant Growth Through Diet and Enteric Health
Acronym: JiVitA-6
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00008000; OPP1163259 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Stunting; Malnutrition; Protein; Enteric Pathogens; Campylobacter Infections
Keywords: linear growth; infant feeding; environmental enteric dysfunction
MeSH Terms: conditions — Growth Disorders; Kwashiorkor; Campylobacter Infections | interventions — Eggs; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: For this 2 x 4 factorial, cluster-randomized trial, 566 previously defined clusters will be assigned independently to 8 different combinations of interventions: 1) azithromycin and protein supplementation; 2) azithromycin and isocaloric supplementation; 3) azithromycin and egg; 4) azithromycin and control (nutrition education); 5) placebo and protein supplementation; 6) placebo and isocaloric supplementation; 7) placebo and egg; 8) placebo and control (nutrition education).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators and outcomes assessors will be blinded to the azithromycin or placebo interventions. Neither participants nor outcomes assessors will be masked to the nutrition interventions. Investigators will be masked to the nutrition interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Placebo & Control (Placebo Comparator): Placebo / Nutrition education
  Interventions: Drug: Placebos; Behavioral: Nutrition Education
- Placebo & Protein Supplement (Experimental): Placebo / Protein-rich blended food / Nutrition education
  Interventions: Drug: Placebos; Dietary Supplement: Protein Supplement; Behavioral: Nutrition Education
- Placebo & Isocaloric Supplement (Placebo Comparator): Placebo / Isocaloric blended food / Nutrition education
  Interventions: Drug: Placebos; Dietary Supplement: Isocaloric Supplement; Behavioral: Nutrition Education
- Placebo & Egg (Experimental): Placebo / Egg / Nutrition education
  Interventions: Drug: Placebos; Dietary Supplement: Egg; Behavioral: Nutrition Education
- Azithromycin & Control (Experimental): Azithromycin / Nutrition education
  Interventions: Drug: Azithromycin Oral Product; Behavioral: Nutrition Education
- Azithromycin & Protein Supplement (Experimental): Azithromycin / Protein-rich blended food / Nutrition education
  Interventions: Drug: Azithromycin Oral Product; Dietary Supplement: Protein Supplement; Behavioral: Nutrition Education
- Azithromycin & Isocaloric Supplement (Experimental): Azithromycin Isocaloric blended food Nutrition education
  Interventions: Drug: Azithromycin Oral Product; Dietary Supplement: Isocaloric Supplement; Behavioral: Nutrition Education
- Azithromycin and Egg (Experimental): Azithromycin Egg Nutrition education
  Interventions: Drug: Azithromycin Oral Product; Dietary Supplement: Egg; Behavioral: Nutrition Education

INTERVENTIONS:
Drug: Azithromycin Oral Product — Azithromycin oral suspension (10 mg/kg; 3 days) administered by study personnel at 6 and 9 months of age
  Other Names: Azithrocin
  Arms: Azithromycin & Control; Azithromycin & Isocaloric Supplement; Azithromycin & Protein Supplement; Azithromycin and Egg
Drug: Placebos — Contain inert excipients only
  Arms: Placebo & Control; Placebo & Egg; Placebo & Isocaloric Supplement; Placebo & Protein Supplement
Dietary Supplement: Protein Supplement — Blended food providing 125 kcal and 10 g protein as egg white powder prepared as porridge and fed daily to infants from 6-12 months of age
  Arms: Azithromycin & Protein Supplement; Placebo & Protein Supplement
Dietary Supplement: Isocaloric Supplement — Blended food providing 125 kcal and 1 g protein as rice powder prepared as porridge and fed daily to infants from 6-12 months of age
  Arms: Azithromycin & Isocaloric Supplement; Placebo & Isocaloric Supplement
Dietary Supplement: Egg — Egg provided daily to infants from 6-12 months of age
  Arms: Azithromycin and Egg; Placebo & Egg
Behavioral: Nutrition Education — Monthly messaging on infant and young child feeding

SUMMARY:
This cluster-randomized controlled trial is designed to address linear growth faltering in 6-12-mo-old Bangladesh infants through a proof-of-concept package of interventions to a) increase intake of high quality protein and b) control enteric pathogens.

DETAILED DESCRIPTION:
Stunting a major public health problem in Bangladesh, where 36% of children under the age of five are too short for their age. While dietary data indicate that protein intakes of infants and young children are largely in line with requirements, the extent to which requirements derived for healthy infants and young children are relevant in the context of frequent infections remains an important research question.

Recent investigations indicate widespread pathogen carriage among Bangladeshi infants, with virtually all having at least one detectable pathogen in nondiarrheal stools by six months of age. Campylobacter and pathogenic E. Coli predominate in this setting. Enteric pathogens can compete with the host for available nutrients or alter nutrient metabolism. Acting via environmental enteric dysfunction, they can alter both digestion-through loss of digestive enzymes-and absorption of nutrients. Microbial translocation may further alter specific amino acid requirements.

Even in the absence of acute diarrheal disease, enteric pathogen carriage is strongly associated with linear growth faltering. Combining the effects of high pathogen burden and poor diet, as indicated by low energy and protein from complementary foods, observational evidence suggests that the potentially preventable length-for-age Z-score deficit may be as high as 0.98.

The present trial will test the combination of a) protein supplementation in the form of a protein-rich blended food or an egg, both fed daily to infants 6-12 months of age, and b) azithromycin treatment for enteric pathogens. The primary outcome will be change in length-for-age Z-score from the 6 to 12 months. Biochemical, microbiological and clinical intermediates will be measured to inform our secondary aims.

ELIGIBILITY:
Inclusion Criteria:

* Born to women enrolled in ongoing community trial (NCT02909179) over a one-year period

Exclusion Criteria:

* Born to women not registered as part of the ongoing community trial (NCT02909179)

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5283 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Length-for-age Z-score (LAZ) at 12 months of age | 12 months

SECONDARY OUTCOMES:
Nutrient biomarkers | 6 and 12 months
  Serum essential, conditionally essential amino acids and choline (by metabolomic analysis); retinol and tocopherols (HPLC); vitamin B12 (microbiological assay); zinc (AAS); ferritin and thyroglobulin (ELISA)
Growth hormone and stress axes biomarkers | 6 and 12 months
  Serum insulin-like growth factor 1 (IGF-1), IGF binding protein 3, cortisol, by ELISA
Enteropathogen burden | 6, 6.5, 9, 9.5, 12, 15, and 18 months
  Campylobacter, enterotoxigenic Escherichia coli (ETEC), enteroaggregative Escherichia coli (EAEC), enteropathogenic Escherichia coli (EPEC), Shigella and Cryptosporidium, by quantitative polymerase chain reaction (qPCR)
Gut microbiota composition | 6, 6.5, 9, 9.5, 12, 15, and 18 months
  Microbial diversity and abundance, by 16S ribosomal RNA sequencing
Environmental enteric dysfunction biomarkers | 6 and 12 months
  Stool myeloperoxidase and intestinal fatty acid-binding protein concentrations and plasma Endogenous endotoxin-core antibody (EndoCAb), by ELISA
Inflammatory biomarkers | 6 and 12 months
  Plasma alpha-1 acid glycoprotein, C-reactive protein and interleukin-6, by ELISA; stool inflammatory cytokines, by ELISA
Bone biomarkers | 6 and 12 months
  Plasma collagen type X and N-Terminal Pro-C-Type Natriuretic Peptide (NT-ProCNP), by ELISA
Morbidity incidence | 6-12 months
  Incident diarrhea/dysentery or respiratory infection, based on weekly recalls
Body composition | 6, 9, 12, 15, and 18 months
  Fat mass by bioelectrical impedence
Antibiotic resistance | 6, 9, 12, 15, and 18 months
  Resistance of commensal E. coli (stool) or S. pneumoniae (nasopharyngeal swab) to panel of antibiotics, by culture

CONTACTS AND LOCATIONS:
Overall Officials: Amanda C Palmer, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Md Iqbal Hossain, PhD, Principal Investigator — International Centre for Diarrhoel Disease Research, Bangladesh
Locations (1):
- JiVitA Maternal and Child & Nutrition Research Site, Gaibandha, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arsenault JE, Brown KH. Dietary Protein Intake in Young Children in Selected Low-Income Countries Is Generally Adequate in Relation to Estimated Requirements for Healthy Children, Except When Complementary Food Intake Is Low. J Nutr. 2017 May;147(5):932-939. doi: 10.3945/jn.116.239657. Epub 2017 Feb 15. PMID 28202639
- [Background] Uauy R. Keynote: rethinking protein. Food Nutr Bull. 2013 Jun;34(2):228-31. doi: 10.1177/156482651303400213. No abstract available. PMID 23964397
- [Background] Lang D; MAL-ED Network Investigators. Opportunities to assess factors contributing to the development of the intestinal microbiota in infants living in developing countries. Microb Ecol Health Dis. 2015 May 29;26:28316. doi: 10.3402/mehd.v26.28316. eCollection 2015. PMID 26031686
- [Background] MAL-ED Network Investigators. Relationship between growth and illness, enteropathogens and dietary intakes in the first 2 years of life: findings from the MAL-ED birth cohort study. BMJ Glob Health. 2017 Dec 28;2(4):e000370. doi: 10.1136/bmjgh-2017-000370. eCollection 2017. PMID 29333282
- [Derived] Palmer AC, Hossain MI, Ali H, Ayesha K, Shaikh S, Islam MT, Johura FT, Pasqualino MM, Rahman H, Haque R, Alland K, Wu LS, Schulze KJ, Chakraborty S, West KP Jr, Alam M, Ahmed T, Labrique AB. Protein supplementation delivered alone or in combination with presumptive azithromycin treatment for enteric pathogens did not improve linear growth in Bangladeshi infants: results of a cluster-randomized controlled trial. Am J Clin Nutr. 2025 Mar;121(3):597-609. doi: 10.1016/j.ajcnut.2024.12.027. Epub 2025 Jan 7. PMID 39788294
- [Derived] Pasqualino MM, Shaikh S, Hossain MI, Islam MT, Ali H, Haque R, Ayesha K, Wu LS, Dyer B, Hasan K, Alland K, Schulze KJ, Johura FT, Alam M, West KP Jr, Ahmed T, Labrique AB, Palmer AC. An Egg Intervention Improves Ponderal But Not Linear Growth Among Infants 6-12 mo of Age in Rural Bangladesh. J Nutr. 2024 Jul;154(7):2290-2299. doi: 10.1016/j.tjnut.2024.05.006. Epub 2024 May 15. PMID 38759886
- [Derived] Tong H, Thorne-Lyman A, Palmer AC, Shaikh S, Ali H, Gao Y, Pasqualino MM, Wu L, Alland K, Schulze K, West KP Jr, Hossain MI, Labrique AB. Prelacteal feeding is not associated with infant size at 3 months in rural Bangladesh: a prospective cohort study. Int Breastfeed J. 2024 Feb 27;19(1):15. doi: 10.1186/s13006-024-00621-4. PMID 38413997